CLINICAL TRIAL: NCT06458972
Title: Safety and Efficacy of Telitacicept in the Treatment of Systemic Lupus Erythematosus (SLE) in the Real World: a Multicenter Retrospective Study
Brief Title: Safety and Efficacy of Telitacicept in the Treatment of Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Jingzhou Central Hospital (Other); Wuhan Central Hospital (Other); Xiangyang Central Hospital (Other); Wuhan No.1 Hospital (Other); China Three Gorges University, Yichang, China (Other); Shanghai Zhongshan Hospital (Other); The First People's Hospital of Jingzhou (Unknown)
Responsible Party: Principal Investigator, Lingli Dong, Professor, Tongji Hospital
Other Study IDs: TJ-IRB20231298
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Telitacicept; adherence; safety; effectiveness
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Systemic lupus erythematosus (SLE) is a highly specific autoimmune disease that involves multiple systems due to abnormal immune activation. It is a classical diffuse connective tissue disease with autoimmune inflammation as its prominent manifestation. B cells are the core of systemic lupus erythematosus (SLE) pathogenesis. B Lymphocyte Stimulator (BLyS, also called BAFF) and A Proliferation-Inducing Ligand (APRIL) are signals for B cell maturation. B Lymphocyte Stimulator (BLyS) participates in promoting the development and maturation of B cells, while A Proliferation-Inducing Ligand (APRIL) participates in promoting the activation of mature B cells and the secretion of antibodies by plasma cells. Telitacicept is composed of the extracellular specific soluble portion of Transmembrane Activator and Calcium-modulating Cyclophilin Ligand (CAML) Interactor (TACI) and the Fragment crystallizable (Fc) segment of human Immunoglobulin G1 (IgG1). It is the only globally approved dual-target biological agent for the treatment of systemic lupus erythematosus (SLE) , blocking B Lymphocyte Stimulator (BLyS) and A Proliferation-Inducing Ligand (APRIL), hindering the development and activation of B cells, and the production of antibodies, comprehensively inhibiting the maturation, proliferation, and differentiation of B cells at different stages. In this study, the investigators will explore the adherence and influencing factors of telitacicept in systemic lupus erythematosus (SLE) patients, its effectiveness, and safety, providing a stronger basis for clinical management of systemic lupus erythematosus (SLE) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, not exceeding 70 years old (including 70 years old);
2. Patients diagnosed with systemic lupus erythematosus (SLE) according to 2019 American College of Rheumatology/European League Against Rheumatism (2019ACR/EULAR) international classification diagnostic criteria;
3. Accepting the treatment of telitacicept.

Exclusion Criteria:

Subjects who meet any of the following criteria should be excluded from this study:

1. Patients with other rheumatic immune system diseases;
2. Patients in the active stage of acute and chronic infections;
3. Patients using other biologics;
4. Patients with wasting diseases such as malignant tumors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic lupus erythematosus (SLE) is a highly specific autoimmune disease involving multiple systems caused by abnormal immune activation. It is a classic diffuse connective tissue disease characterized by autoimmune inflammation. Our study population is the people who confirmed diagnosis of systemic lupus erythematosus (SLE) by 2019 American College of Rheumatology/European League Against Rheumatism (2019ACR/EULAR) International classification diagnostic criteria and patients receiving Tacrolimus injections.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Estrogens in Lupus National Assessment-Systemic Lupus Erythematosus Disease Activity Index （SELENA-SLEDAI） | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Safety of Estrogens in Lupus National Assessment-Systemic Lupus Erythematosus Disease Activity Index （SELENA-SLEDAI） is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with SLE. It is scored by a table named "SELENA-SLEDAI (Systemic Lupus Erythematosus Disease Activity Index) INSTRUMENT SCORE" . The minimum and maximum values are 0 points and 105 points separately, but very few patients score higher than 45 points. Higher scores indicate higher disease activity.
Physician's Global Assessment | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Physician's global assessment for patients with Systemic Lupus Erythematosus (SLE) is a subjective assessment tool used by a same physicians to evaluate the overall disease activity based on clinical observations and patient reports(the patient's symptoms, physical examination findings, laboratory results, and any other relevant clinical information). The physician's global assessment (PGA) scale typically ranges from 0 to 3, with 0 representing no disease activity and 3 representing severe disease activity. Some variations of the scale may include intermediate markers, such as 1 and 2, to indicate varying degrees of disease activity.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline and Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a questionnaire-based tool (FACIT-F, Vision 4) used to measure fatigue in patients. It consists of multiple items, each focusing on a different aspect of fatigue. The items are typically rated on a scale from 0 to 4, with 0 representing "not at all" and 4 representing "very much". Example items include: "I feel tired" or "I'm too tired to working". Higher scores indicate less fatigue.
Serum anti-double stranded DNA (anti-dsDNA) | Baseline, Month 6, Month 12 after injecting Telitacecipt
  to describe the qualitative feature of systemic lupus erythematosus (SLE) patients' serum anti-double stranded DNA (anti-dsDNA).
Serum complement C3 levels | Baseline, Month 6, Month 12 after injecting Telitacecipt
  Serum complement C3 levels (g/L)
Serum complement C4 levels | Baseline, Month 6, Month 12 after injecting Telitacecipt
  Serum complement C4 levels (g/L)
Serum immunoglobulin quantification | Baseline, Month 6, Month 12 after injecting Telitacecipt
  Serum immunoglobulin quantification (g/L)
Levels of C-reactive protein (CRP) levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of C-reactive protein (CRP) levels (mg/L)
Levels of interleukin-10 (IL-10) levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of interleukin-10 (IL-10) levels (pg/mL)
Levels of ferritin levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of ferritin levels (ug/L)
the safety of telitacicept for SLE patients | Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  The probability of adverse reactions （Local adverse reactions after injection） and the probability of major drug-related adverse events
the reasons for medication discontinuation | Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  The investigators will survey the reasons for medication discontinuation by telephone or outpatient follow-up ,the different reasons include economic reasons、 disease improved or be a stable condition、 poor effect、 arise adverse reaction, etc.
Levels of leukocyte levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of leukocyte levels （*10^9/L）
Levels of hemoglobin (Hb) levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of hemoglobin (Hb) levels (g/L)
Levels of blood platelet (PLT) levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of blood platelet (PLT) levels (*10^9/L)
routine urine test | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  To evaluate the grade of urine occult blood and urine protein
Levels of erythrocyte sedimentation rate (ESR) levels | Baseline and Month1, Month 2, Month 3, Month 6, Month 9, Month 12 after injecting Telitacecipt
  Levels of erythrocyte sedimentation rate (ESR) levels (mm/h）
Levels of interleukin-6 (IL-6) levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of interleukin-6 (IL-6) levels (pg/mL)
Levels of interleukin-4 (IL-4) levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of interleukin-4 (IL-4) levels (pg/mL)
Levels of interleukin-2 (IL-2) levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of interleukin-2 (IL-2) levels (pg/mL)
Levels of tumor necrosis factor-α (TNF-α) levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of tumor necrosis factor-α (TNF-α) levels (pg/mL)
Levels of interferon-γ（IFN-γ） levels | Baseline and Month 6，Month 12 after injecting Telitacecipt
  Levels of interferon-γ（IFN-γ） levels (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Lingli, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China